CLINICAL TRIAL: NCT03083925
Title: Viatorr Control Expansion Compared to Bare-metal and Regular Viatorr for Complications of Portal Hypertension
Brief Title: Viatorr CX Case-control Study for Complications of Portal Hypertension
Acronym: VIATORR-CX
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Jonel Trebicka, Prof. Dr., University Hospital, Bonn
Other Study IDs: TIPS-CX
Record Dates: First submitted 2017-03-03; First posted 2017-03-20 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Liver Cirrhoses; Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, stool, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bare metal stent (BMS) TIPS: retrospective patients receiving BMS-TIPS for treatment of complications of portal hypertension.
  Interventions: Device: TIPS
- Regular Viatorr (RV) TIPS: retrospective patients receiving RV-TIPS for treatment of complications of portal hypertension.
  Interventions: Device: TIPS
- Viatorr Control Expansion (VCX)TIPS: prospective patients receiving VCX-TIPS for treatment of complications of portal hypertension.
  Interventions: Device: TIPS

INTERVENTIONS:
Device: TIPS — Transjugular Intrahepatic Portosystemic Shunt

SUMMARY:
To evaluate the clinical benefits in the patients receiving Viatorr CX over a period of 12 months of structured Follow-up (before TIPS, at TIPS, 1 week after TIPS, at 6 weeks, 4 months, 6 months, 9 months, 12 months), regarding clinical endpoints, such as HE, readmission, liver injury, cardiac function, response to TIPS and the passive expansion of the stents in real life.

DETAILED DESCRIPTION:
Case-control study using the patients in the University Clinic Bonn receiving Viatorr CX (n=40), using a comparison ration 1:1:1 to Viatorr and bare metal stents.

Of these patients, 20 patients will receive Viatorr CX and the assessement of the width of the stent as outlined in the JVIR-paper published this year.

The Viatorr and BMS controls with similar age, gender, Child, MELD and indication for TIPS.

A total of 125 patients with the primary composite-endpoint HE/readmission will be investigated Secondary endpoints are liver injury, cardiac function, response to TIPS and the passive expansion of the stents in real life.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for TIPS

Exclusion Criteria:

* Contraindication for TIPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case-control study using the patients in our center receiving Viatorr CX (n=40), using a comparison ration 1:1:1 to Viatorr and bare metal stents (all available data from our center). Thereby, we will choose 20 patients receiving Viatorr CX and the assessement of the width of the stent as outlined in the JVIR-paper published this year. The Viatorr and BMS controls with similar age, gender, Child, MELD and indication for TIPS. We will investigate a total 125 patients with the primary composite-endpoint HE/readmission, and secondary endpoints will be liver injury, cardiac function, response to TIPS and the passive expansion of the stents in real life.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Readmissions | 12 months
  Number of readmissions will be documented using a structured CRF

SECONDARY OUTCOMES:
Hepatic encephalopathy (HE) | 12 months
  Number of Episodes of overt HE (West Haven Criteria > Grad I)
Liver injury | 12 months
  Increase in liver function tests
Response to TIPS | 12 months
  grade of ascites after TIPS

CONTACTS AND LOCATIONS:
Overall Officials: Jonel Trebicka, MD, PhD, Principal Investigator — Laboratory for Liver Fibrosis and Portal Hypertension
Locations (1):
- Laboratory for Liver Fibrosis and Portal Hypertension, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No